CLINICAL TRIAL: NCT04788784
Title: Mixed-method Study to Evaluate Acceptability, Perceived Toxicity, Preference and Health-related Quality of Life Among HIV Patients Switching to a Dual Therapy Such as the Dovato Regimen
Brief Title: Patient-Reported Outcomes HIV BItherapy
Acronym: PROBI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Paris 7 - Denis Diderot (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Dr Martin Duracinsky, Doctor, University Paris 7 - Denis Diderot
Other Study IDs: PROBI
Record Dates: First submitted 2021-03-02; First posted 2021-03-09 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: HIV/AIDS and Infections; Patient Preference
Keywords: HIV dual therapy; Patient-reported Outcomes; Health-Related Quality of Life
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections; Patient Preference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
HIV Treatment simplification strategies that involve switching cART regimens from four or three antiretrovirals to two in virologically suppressed patients living with HIV are now available in order to reduce long-term toxicity and enhance treatment adherence. Dolutegravir is a second-generation integrase strand transfer inhibitor (INSTI) with noticeable advantages, including a high genetic barrier to drug resistance, once-daily dosing and lower risk of drug-drug interactions because this agent does not inhibit or induce cytochrome P450 isoenzymes or P-glycoprotein transporters. Dolutegravir is generally well tolerated and the INSTI class is considered to be more "metabolically friendly" compared with other drug classes such as protease inhibitors (PIs). Thus, the combination of dolutegravir plus a second active agent is a particularly inviting option for maintenance treatment and research in this area is evolving. However, though safety and efficacy of dolutegravir are well known, there is no study evaluating patient-reported outcomes (PROs), i.e. subjective and self-reported measures of the patient's health perception. In an era of the efficacy of HIV regimens are more and more comparable, the main discriminant criteria to choose the best treatment option are now adherence and self-reported measures of a patient's health - termed "patient-reported outcomes" (PROs).

The study, based on a mixed methodology, include a qualitative part and a quantitative part. The qualitative study will explore patients' and health care professionals' perceptions, knowledge, and representations of triple or quadruple and dual therapies and detect the degree of agreement or disagreement between patients' and practitioners' perspectives. The quantitative study's main objective is to measure the Dovato regimen's impact on a patient's perception (Patient-Reported Outcomes - PRO) on acceptability, toxicity, preference, and Health-Related Quality of Life (HRQL). PRO are collected through self-administered questionnaires at D0 (when the patient switch treatment), M1 and M6.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected by HIV-1
* Patients who are prescribed the Dovato regimen by their clinicians in routine care
* Patients previously under the cART regimen with three or four antiretrovirals
* HIV-RNA <=50 copies/mL for at least 3 months
* 18 years old and more
* Ability to understand and respond to questionnaires

Exclusion Criteria:

* Pregnant or breastfeeding women
* Known hypersensitivity to dolutegravir and lamivudine, their metabolites or formulation excipient
* Active, serious infection (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to inclusion
* Any other clinical condition or prior therapy that, in the investigator's opinion, would make the subject unsuitable for the study, or unable to comply with protocol requirements.
* Active CDC Category C disease
* Treatment with radiation therapy, cytotoxic chemotherapeutic agents 30 days before inclusion
* Patient co-infected with HBV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1 patients who are prescribed a Dovato regimen by their clinicians in routine care for any reason. The patient must be able to read in order to fill up the questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Change of the patient perception (Patient-Reported Outcomes - PRO) after a switch from HIV tritherapy to DOVATO dual therapy on the perceived toxicity of the treatment. | Day 0, Month 1 and Month 6
  A score of perceived toxicity and preference: measured by the scale developed during a previous qualitative step of the study (PTP scale) on the day of the switch, 1 month after the switch and 6 month after the switch.
Change of the patient perception (Patient-Reported Outcomes - PRO) after a switch from HIV tritherapy to DOVATO dual therapy on the acceptability of the treatment. | Day 0, Month 1 and Month 6
  A score of acceptability (at baseline only): measured by the scale developed during a previous qualitative step of the study (Acceptability scale) on the day of the switch, 1 month after the switch and 6 month after the switch.
Change of the patient perception (Patient-Reported Outcomes - PRO) after the switch from HIV tritherapy to DOVATO dual therapy on Health-Related Quality of Life (HRQL) | Day 0, Month 1 and Month 6
  The treatment impact (TI, 10) dimension of the PROQOL-HIV questionnaire will measure HRQL on the day of the switch, 1 month after the switch and 6 month after the switch.

SECONDARY OUTCOMES:
Change of the patient perception (Patient-Reported Outcomes - PRO) after the switch from HIV tritherapy to DOVATO dual therapy on the percieved HIV symptoms | Day 0, Month 1 and Month 6
  HIV Symptom Index, a 20 items index on different symptoms experienced by HIV patients on the day of the switch, 1 month after the switch and 6 month after the switch.
Change of the patient perception (Patient-Reported Outcomes - PRO) after the switch from HIV tritherapy to DOVATO dual therapy on adherence with the dual therapy | Day 0, Month 1 and Month 6
  Adherence ANRS (Agence nationale de recherches sur le sida et les hépatites virales - French agency for AIDS and viral hepatitis research) questionnaire of 3 items
Factors associated with high preference versus low preference for dual therapy | Day 0, Month 1 and Month 6
  Describe the factors associated with high acceptability of Dovato regimen (acceptability scale)
Efficacy of the Dovato regimen through Week 24 | Day 0, Month 1 and Month 6
  Percentage of Participants With Human Immunodeficiency Virus-1 (HIV-1) RNA <50 Copies (c)/Millilitre (mL) Through Week 24
Kinetic of CD4 through Week 24 | Day 0, Month 1 and Month 6
  Change From Baseline in Cluster of Differentiation (CD)4+ Cell Counts Over Time

CONTACTS AND LOCATIONS:
Overall Officials: Martin Duracinsky, PhD, Principal Investigator — URC-ECO, AP-HP & UMR 1123, Université de Paris, Inserm
Locations (3):
- France (3):
  - Hôpital de Bicêtre, Le Kremlin-Bicêtre
  - Centre hospitalier de Cornouaille, Quimper
  - Centre Hospitalier de Saint-Denis - Hôpital Delafontaine, Saint-Denis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duracinsky M, Alain T, Zucman D, Rousset Torrente O, Brown Hajdukova E, Hocqueloux L, Allavena C, Marcellin F, Chassany O. Patient-reported outcomes among people living with HIV switching to dual therapy with dolutegravir/lamivudine: results from the PROBI study. Ther Adv Infect Dis. 2025 Oct 14;12:20499361251321728. doi: 10.1177/20499361251321728. eCollection 2025 Jan-Dec. PMID 41112057
- [Derived] Alain T, Marcellin F, Bessonneau P, Hocqueloux L, Muehlan H, Allavena C, Zucman D, Villalong-Olives E, Chassany O, Duracinsky M. Sex Differences in Patient-Reported Outcomes Among People Living With HIV Switching to an Oral Dual Therapy: Results From the PROBI Study. AIDS Res Treat. 2025 Oct 2;2025:1850783. doi: 10.1155/arat/1850783. eCollection 2025. PMID 41078979